CLINICAL TRIAL: NCT06228638
Title: CognivAiD Real-World Evidence Clinical Registry
Brief Title: CognivAiD Real-World Evidence Clinical Registry (CONNECT Registry)
Acronym: CONNECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moleac Pte Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAFE2022_01
Record Dates: First submitted 2024-01-15; First posted 2024-01-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Memory Impairment; Dementia, Vascular
Keywords: CognivAiD; Memory Cognitive Impairment; Vascular Dementia; Traditional Chinese Medicine
MeSH Terms: conditions — Memory Disorders; Dementia, Vascular | interventions — sailuotong

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CognivAID (Sailuotong) — CognivAiD is 27.27 mg of panax ginseng standard extract, 27.27 mg of gingo biloba standard extract and 5.46 mg of crocus sativus standard extract which is equal to 60mg /capsule .CognivAiD is available at 60 mg /cap 2 caps twice a day.
  Other Names: SAILUOTONG

SUMMARY:
This is an observational, prospective cohort of patients who were prescribed or have taken CognivAiD as prescribed by the attending physician. The safety and efficacy of CognivAiD have been established in clinical studies. The registry will assess the safe use and effectiveness of CognivAiD in a real-world setting. The registry is designed as a product registry in clinical practice. The design also takes into account the different scenarios of product use in the real world (e.g., switching therapies during follow-up, use of multiple products in combination or sequence, different dosing, and compliance).

DETAILED DESCRIPTION:
While the safety and efficacy of CognivAiD is established in clinical studies, this registry will assess the safe use and effectiveness of CognivAiD in the real-world setting. The design also takes into account the different scenarios of product use in the real world (e.g., switching therapies duObjectivesThe primary objective of this registry is to evaluate the use, safety, and effectiveness of CognivAiD This project is not a clinical trial wherein an active intervention intended to change human subject's outcome is implemented and takes decision-making away from the physician and patient. This registry uses an observational study design that does not specify or assign treatments or therapies. The registry is designed by keeping as closely as possible to real-world practice and as unobtrusive as possible to closely reflect usual practice and normal standards of care.

There are few inclusion and exclusion criteria to include a broad range of participants to make the results more generalizable. Participants are observed as they present for care and the data collected reflects existing tests, measurements, and treatments a healthcare provider customarily uses. Participation in the registry is entirely voluntary.

The primary objective of the registry is to evaluate the use, safety, and effectiveness of CognivAiD in a real-world setting. The primary data elements include the reporting of side effects and adverse events. Data collection and includes demographics, education, number of years, past medical history, CognivAiD information and, neurological status by the standard clinical practice and normal standard of care. Cognitive Assessment will be performed as per routine clinical visit. Collected data will be entered into the online study database.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Legal age as per country requirement
* Already taking or having to receive a prescription for CognivAiD (decision must have been made before consideration to participate in the registry)
* Agrees to be included in the registry, provides written consent inclusion criteria
* Male or female
* Legal age as per country requirement
* Already taking or having to receive a prescription for CognivAiD (decision must have been made before consideration to participate in the registry)
* Agrees to be included in the registry, provides written consent, and allows retrieval and analysis of data by local requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population would involve patients with MCI, Vascular dementia, Dementia who are taking or prescribed CognivAiD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety reporting | baseline, one month, 3rd month, 6th month, 9th month and one year
  The Registry will collect adverse events or side effects reported by the doctors .

CONTACTS AND LOCATIONS:
Overall Officials: Narayanaswamy U Venketasubramanian, MD, Principal Investigator — Raffles Hospital
Locations (1):
- Raffles Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share unidentified data with other investigators who are part of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: one year

REFERENCES:
- [Result] Zhang Y, Lin L, Liu GY, Liu JX, Li T. [Pharmacokinetics and brain distribution of ginsenosides after administration of sailuotong]. Zhongguo Zhong Yao Za Zhi. 2014 Jan;39(2):316-21. Chinese. PMID 24761653
- [Result] Seto SW, Chang D, Ko WM, Zhou X, Kiat H, Bensoussan A, Lee SM, Hoi MP, Steiner GZ, Liu J. Sailuotong Prevents Hydrogen Peroxide (H(2)O(2))-Induced Injury in EA.hy926 Cells. Int J Mol Sci. 2017 Jan 5;18(1):95. doi: 10.3390/ijms18010095. PMID 28067784
- [Result] Zhang Y, Liu J, Yao M, Song W, Zheng Y, Xu L, Sun M, Yang B, Bensoussan A, Chang D, Li H. Sailuotong Capsule Prevents the Cerebral Ischaemia-Induced Neuroinflammation and Impairment of Recognition Memory through Inhibition of LCN2 Expression. Oxid Med Cell Longev. 2019 Sep 3;2019:8416105. doi: 10.1155/2019/8416105. eCollection 2019. PMID 31565154
- [Result] Steiner GZ, Yeung A, Liu JX, Camfield DA, Blasio FM, Pipingas A, Scholey AB, Stough C, Chang DH. The effect of Sailuotong (SLT) on neurocognitive and cardiovascular function in healthy adults: a randomised, double-blind, placebo controlled crossover pilot trial. BMC Complement Altern Med. 2016 Jan 13;16:15. doi: 10.1186/s12906-016-0989-0. PMID 26762282
- [Result] Chang D, Liu J, Bilinski K, Xu L, Steiner GZ, Seto SW, Bensoussan A. Herbal Medicine for the Treatment of Vascular Dementia: An Overview of Scientific Evidence. Evid Based Complement Alternat Med. 2016;2016:7293626. doi: 10.1155/2016/7293626. Epub 2016 Dec 27. PMID 28115971